CLINICAL TRIAL: NCT02426502
Title: Once Daily Dosing to Improve Medication Adherence and Patient Satisfaction in Kidney Transplant Recipients: A Pilot Study
Brief Title: Once Daily Dosing to Improve Medication Adherence and Patient Satisfaction in Kidney Transplant Recipients
Acronym: OnceDaily
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Astellas Pharma Canada, Inc. (Industry)
Responsible Party: Principal Investigator, John Gill, Assistant Professor, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H14-01441
Record Dates: First submitted 2015-04-08; First posted 2015-04-27 (Estimated); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: End-Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Tacrolimus; Cyclosporine; Mycophenolic Acid; Azathioprine; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Conversion to once daily dosing (Experimental): The conversion to a once daily dosing regimen will be accomplished in three phases (1-conversion to Advagraf; 2-conversion of non-immunosuppressant drugs and; 3-conversion of patients taking twice daily MPA to once daily MPA). No control group.
  Interventions: Drug: Conversion to Advagraf; Drug: conversion of non-immunosuppressant drugs to once daily; Drug: Conversion to once daily MPA

INTERVENTIONS:
Drug: Conversion to Advagraf — Prograf treated patients will convert to Advagraf using a 1: 1 conversion for a period of one week. The dose will then be titrated based on tacrolimus trough levels obtained 7 days after conversion. Cyclosporine (Neoral) treated patients will initiate Advagraf 0.075 mg/kg/day, 24 hours after their last cyclosporine dose. Participants will be provided with Advagraf and instructed how to start this new medication
  Other Names: Prograf, Cyclosporine (Neoral), Advagraf
Drug: conversion of non-immunosuppressant drugs to once daily — * Conversion of anti-hypertensive medications: converted to once daily alternatives with the goal of maintaining blood pressure at the same or lower level prior to conversion.
  * Conversion of all other medications: changed to once daily formulations of the same medication or a once daily alternative.
  Other Names: anti-hypertensive medications, non-immunosuppressant drugs
Drug: Conversion to once daily MPA — * Conversion to once daily MPA: Patients taking mycophenolate mofetil (MMF) will receive 1.0 gram once daily, while patients receiving Myfortic will receive 720 mg once daily.
  * Conversion to once daily Myfortic: Patients prescribed proton pump inhibitors (PPIs) and MMF will be switched to equivalent dose Myfortic for a period of one month prior to conversion to once daily MPA.
  * Patients taking azathioprine will be maintained on the same dose.
  * Patients will be maintained on the same prednisone dose.
  Other Names: Mycophenolate Mofetil, Myfortic, Azathioprine, Prednisone

SUMMARY:
Patient failure to take medications as prescribed (medication non-adherence) is now identified as an important cause of kidney transplant failure. The availability of new drugs that are taken once daily may improve patient adherence compared to older drugs that had to be taken twice per day. In this study, patients will be converted to a medication schedule where all medications are taken once daily with the goal of improving patient adherence and satisfaction.

DETAILED DESCRIPTION:
The current pilot study will first demonstrate the safety and feasibility of converting maintenance transplant recipients to a once daily regimen, while measure of patient satisfaction and adherence are secondary outcomes. The purpose of this study is to determine the safety and feasibility of converting maintenance kidney transplant recipients (i.e. those more than one year post transplantation) to a once daily drug regimen (including immunosuppressant and non-immunosuppressant drugs). We believe that conversion to a once daily (O.D.) medication regimen for both immunosuppressive and non-immunosuppressive medications will be associated with increased patient adherence and satisfaction.

Immunosuppressant non-adherence is considered the leading potentially avoidable cause of allograft failure, with non-adherent patients having a seven fold higher odds of graft failure than adherent patients. Although medication non-adherence is multi-factorial, simplification of medication requirements has been associated with improved adherence in the non-transplant setting.

There are few prospective studies examining strategies to improve immunosuppressant adherence. The proposed study has significant potential to improve medication adherence and satisfaction in kidney transplant recipients which may ultimately lead to an improvement in long-term outcomes.

The major barrier to establishing a once daily medication regimen in maintenance kidney transplant recipients (i.e. patients ≥ 12 months post transplantation) was related to the requirement to prescribe calcineurin inhibitors twice daily. The development of Advagraf (tacrolimus extended release capsules), which is approved for prevention of rejection in kidney transplant recipients, now provides an opportunity to convert patients to a once daily immunosuppressant medication regimen.

The other maintenance immunosuppressant medications used in kidney transplantation are Mycophenolic acid (MPA), azathioprine and prednisone.

Mycophenolic acid (MPA) was first made available for use in kidney transplantation in 1995 in the form of the prodrug mycophenolate mofetil (MMF); this was later followed by the introduction of mycophenolate sodium (Myfortic).

The recommended dose of MMF and Myfortic are 2g/day and 1440 mg/day respectively in de novo transplant recipients. In clinical practice, maintenance patients (i.e. those who are more than 1 year post transplantation) are often not maintained on the recommended initial (see below). In studies involving patients prescribed the recommended initial daily dose, MPA exposure is highly variable: The 12 hour area under the curve (AUC) ranges anywhere between 15 and 115 mg*h/L. In the first post transplant year, a 12 hour AUC of 30 -60 mg*h/l is recommended based on studies showing an increased incidence of rejection when the AUC < 30 mg*h/l, and no additional efficacy benefit with AUC > 60 mg*h/l in cyclosporine treated patients.

A relationship between MPA exposure and acute rejection beyond 3 months has not been demonstrated. There is a paucity of studies examining the concentration-effect relationship beyond the first post transplant year and thus there are no established recommendations for MPA exposure after the first post-transplant year. In clinical practice a significant proportion of long-term (≥ 1 year post transplant) MPA treated patients will be prescribed less than the recommended dose of MPA due to a variety of reasons including patient intolerance (usually gastrointestinal or hematological). Most reductions in MPA dose are undertaken in the first few months after transplantation when renal allograft dysfunction or hypoalbuminemia may have increased free MPA exposure and possibly increased drug related side effects. Importantly recent controlled studies in both de novo and maintenance transplant patients have demonstrated the safety of once daily MPA dosing using less than the initial recommended daily dose.

Prednisone may or may not be prescribed in maintenance transplant recipients. Maintenance prednisone dose varies between 5 -10 mg once daily or every other day.

Azathioprine is an established once daily medication.

A significant criticism of one daily immunosuppressant regimens has been that patients will still be required to take other medications multiple times per day. Uniquely the proposed study will convert all medications (immunosuppressant and non-immunosuppressants) to a once daily regimen.

In summary, advances in immunosuppressant drugs now make it possible to consider a once daily immunosuppressant regimen in maintenance kidney transplant recipients.

Eligible patients will be screened and consented at the hospital by the study team. The conversion to a once daily dosing regimen will be accomplished in three phases: 1) conversion to Advagraf; 2) conversion of non-immunosuppressant drugs and; 3) conversion of patients taking twice daily MPA to once daily MPA.

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric patients (≥ 12 years) and adult ≥ 18 years
2. Kidney only transplant recipients ≥ 12 months post transplantation
3. Patients prescribed calcineurin inhibitor in the form of tacrolimus, cyclosporin and/or Advagraf
4. Patients without a PRA who have only had one transplant and are deemed clinically low risk by the principle investigator prior to approach.
5. Patients prescribed ≤ 1.0 gram/day of mycophenolate mofetil or ≤ 720 mg/day of mycophenolate sodium continuously in the 3 months prior to the start of the study, or patients prescribed higher doses of these drugs but taking less than the prescribed dose
6. Patients prescribed azathioprine instead of mycophenolate mofetil or mycophenolate sodium, or patients not prescribed any of these drugs.

Inclusion Criteria at British Columbia Children's Hospital:

1. Pediatric patients ≥ 14 years old. Although the protocol has an inclusion criteria of pediatric patients of ≥ 12 years of age, we will only be approaching those ≥ 14.
2. Kidney transplant recipient of ≥ 12 months post transplantation.

Exclusion Criteria:

1. Unable to provide informed consent
2. Patients who previously underwent desensitization for Human Leukocyte Antigen (HLA) or ABO incompatibility
3. Patients with a Panel Reactive Antibody (PRA) ≥ 30% prior to transplantation
4. Participation in another interventional study
5. Glomerular Filtration Rate (GFR)< 25 ml/min/1.73m2
6. Unstable allograft function defined by any of the following:

   i) Acute rejection within the preceding 6 months ii) Biopsy proven chronic humoral rejection at any time iii) Presence of donor specific antibodies at any time prior to or after transplantation iv) Biopsy evidence of de novo or recurrent glomerular disease v) Patients with evidence of declining kidney function (drop in estimated GFR ≥ 5 ml/min/1.73m2 in the previous year)
7. Pregnancy or planned pregnancy in the next 12 months (Note: participants for the study are transplant recipients and will be aware of the inability to become pregnant while prescribed MPA. We will confirm the patient is not pregnant and not planning to become pregnant as part of screening).
8. Patients otherwise considered medically unsuitable for enrolment by their treating physician including previous history of non-adherence.
9. Active infection or treatment for chronic infection (for example active cytomegalovirus, polyoma virus, hepatitis B or C infection, HIV).
10. Active malignancy (excluding non-melanoma skin cancer)
11. Patients in whom conversion to a once daily medication regimen is not feasible because of polypharmacy.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2016-04; Primary Completion 2022-08-10 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients not meeting safety criteria | 1 year after enrollment of the twenty-fifth participant
  Progression between phases will be based on assessment of safety. Patients not meeting safety criteria will not be able to progress between stages and will be withdrawn from the study.
Feasibility: Number of patients successfully converted to a once daily dosing regimen | 12 months
  The proportion of patients that can successfully be converted to a once daily regimen
Feasibility: Number of patients successfully converted to a once daily dosing regimen | Up to 2 years
  The proportion of patients that can successfully be converted to a once daily regimen

SECONDARY OUTCOMES:
Patient Adherence to Dosing Regimen | Baseline
  Adherence will be assessed by the Basel assessment of adherence to immunosuppressive medications scale (BAASIS)
Patient Adherence to Dosing Regimen | Baseline
  Adherence will be assessed by the percent coefficient of variation in calcineurin inhibitor drug levels.
Patient Adherence to Dosing Regimen | 12 months
  Adherence will be assessed by the Basel assessment of adherence to immunosuppressive medications scale (BAASIS)
Patient Adherence to Dosing Regimen | 12 months
  Adherence will be assessed by the percent coefficient of variation in calcineurin inhibitor drug levels.
Patient Adherence to Dosing Regimen | 24 months
  Adherence will be assessed by the percent coefficient of variation in calcineurin inhibitor drug levels.
Patient Adherence to Dosing Regimen | 24 months
  Adherence will be assessed by the Basel assessment of adherence to immunosuppressive medications scale (BAASIS)
Patient Satisfaction | Baseline
  Patient satisfaction will be assessed by survey
Patient Satisfaction | 12 months
  Patient satisfaction will be assessed by survey
Patient Satisfaction | 24 months
  Patient satisfaction will be assessed by survey

CONTACTS AND LOCATIONS:
Overall Officials: John Gill, MD, Principal Investigator — St. Paul's Hospital
Locations (3):
- Canada (3):
  - BC Children Hospital, Vancouver, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia